CLINICAL TRIAL: NCT06467409
Title: A Multicenter, Randomized, Double-blind, Placebo, Positive Drug Parallel Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of LPM3480392 Injection for Moderate to Severe Pain After Orthopedic Surgery
Brief Title: Phase II Clinical Trial to Evaluate the Efficacy and Safety of LPM3480392 Injection for Moderate to Severe Pain After Orthopedic Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LY03014/CT-CHN-204
Record Dates: First submitted 2024-01-26; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- morphine hydrochloride injection (Active Comparator)
  Interventions: Drug: morphine hydrochloride injection
- LPM3480392 injection group 1 (Experimental)
  Interventions: Drug: LPM3480392 Injection
- LPM3480392 injection group 2 (Experimental)
  Interventions: Drug: LPM3480392 Injection
- LPM3480392 injection group 3 (Experimental)
  Interventions: Drug: LPM3480392 Injection
- LPM3480392 injection group4 (Experimental)
  Interventions: Drug: LPM3480392 Injection

INTERVENTIONS:
Drug: Placebo — patient-controlled analgesia(PCA) administration
  Arms: Placebo
Drug: morphine hydrochloride injection — patient-controlled analgesia(PCA) administration
  Arms: morphine hydrochloride injection
Drug: LPM3480392 Injection — patient-controlled analgesia(PCA) administration
  Arms: LPM3480392 injection group 1
Drug: LPM3480392 Injection — patient-controlled analgesia(PCA) administration
  Arms: LPM3480392 injection group 2
Drug: LPM3480392 Injection — patient-controlled analgesia(PCA) administration
  Arms: LPM3480392 injection group 3
Drug: LPM3480392 Injection — patient-controlled analgesia(PCA) administration
  Arms: LPM3480392 injection group4

SUMMARY:
A randomized, double-blind, placebo/positive drug parallel controlled design was used to evaluate the preliminary efficacy and safety of intravenous infusion of LPM3480392 injection using different dosing regimens in subjects with moderate to severe pain after Orthopedic surgery

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent form (ICF) and comply with the trial procedures before starting the trial-related activities;
2. Over 18 years old , male or female;
3. Body mass index (BMI) 18-28 kg/m2 (including the boundary value)；
4. Subjects who plan to undergo unilateral total knee replacement or unilateral knee ligament reconstruction under general anesthesia; ;
5. American Society of Anesthesiologists(ASA )grade I ~ II;
6. Female subjects with a negative pregnancy test at Screening. Male and female subjects agree to take effective contraceptive measures throughout the study and for at least 1 month after medication;
7. the numerical rating scale(NRS) score at rest was ≥ 4 points within 4 hours after surgery.

Exclusion Criteria:

1. Known history of allergy to any component of the investigational product, or allergy or contraindication to the anesthetic/analgesic drugs used in the study;
2. Had any of the following conditions or medical history:

   1. History of stroke, cognitive dysfunction, or epilepsy (excluding convulsions caused by previous febrile convulsions in children);
   2. History of difficult airway, such as obstructive sleep apnea syndrome, bronchial asthma, chronic respiratory diseases or other serious respiratory diseases;
   3. Subjects with a history of myocardial infarction, angina pectoris, severe arrhythmia of degree II or above atrioventricular block, or New York Heart Association(NYHA) Class II or above within 6 months prior to screening;
   4. History of vestibular dysfunction or motion sickness;
   5. Have a history of diabetes and glycosylated hemoglobin ≥ 9% during the screening period;
   6. Esophagitis;
   7. Paralytic gastrointestinal obstruction;
   8. The presence of other acute and chronic pain conditions preoperatively or in combination with other bodily pain conditions that confound the evaluation of postoperative pain.
3. Medications affecting postoperative analgesia before randomization ：

   a) Opioid analgesics taken continuously for more than 10 days for any reason within 3 months prior to randomization, or taking drugs that involving analgesia prior to randomization and The time from last drug use to randomization is less than 5 half-lives( in accord with label ; unless t1/2 is unkown，execute according to 48h ) ,including but not limited to: ketamine, non-steroidal anti-inflammatory drugs (aspirin, acetaminophen, indomethacin, diclofenac, ibuprofen, parecoxib sodium, etc.), alpha adrenoceptor agonists (dexmedetomidine hydrochloride, clonidine, etc.), glucocorticoids (dexamethasone hydrochloride, hydrocortisone, methylprednisolone, etc., except for topical or topical use of glucocorticoids), antiepileptic drugs (carbamazepine, sodium valproate, etc.), sedative drugs (diazepam, estazolam, midazolam, alprazolam, barbiturate, phenobarbital and chloral hydrate, etc.); b. Use of Chinese herbal medicine or Chinese patent medicine which has the function of analgesia, sedation, antiemetic within 48h prior to randomization.
4. Systolic blood pressure less than 90 mmHg or greater than 160 mmHg and diastolic blood pressure 60 mmHg or greater in screening phase;
5. oxygen saturation by pulse oximetry(SpO2) < 92% at screening ;
6. Corrected QT interval(QTc )> 450 ms for males and > 460 m for females at screening ;
7. Patients with abnormal liver and kidney function during screening period:alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 1.5 times of normal value, total bilirubin higher than the upper limit of normal value, serum creatinine (Cr) > 1.5 times of the upper limit of normal value during screening period;
8. Subjects with coagulation abnormalities (PT prolonged more than 3 seconds above the upper limit of normal and/or activated partial thromboplastin time(APTT) prolonged more than 10 seconds above the upper limit of normal) during the screening period; and the investigator confirmed that the abnormalities were clinically significant;
9. History of drug abuse or drug abuse before screening;
10. Positive result in screening of drugs of abuse via urinalysis;
11. Lactating mothers;
12. hepatitis C virus (HCV) antibody, treponema pallidum antibody, human immunodeficiency virus (HIV) antibody positive ;
13. Participation in any medication (excluding vitamins and minerals) within 3 months prior to informed consent Quality) Clinical trial personnel, except for those not using investigational drugs;
14. subjects who are judged by the investigator to be not suitable for this clinical trial, including but not limited to the presence of conditions that may confound the interpretation of efficacy, safety, or tolerability data in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
SPID48 | 48 hours
  the Sum of Pain Intensity Differences in Pain Score from baseline Over 48 Hours

SECONDARY OUTCOMES:
Cumulative dose of rescue analgesic drugs | 48 hours
Incidence of adverse events | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China